CLINICAL TRIAL: NCT01146340
Title: Phase I/II Study of Dose-Escalated Hypofractionated Radiotherapy for Low- and Intermediate-Risk Prostate Cancer
Brief Title: Safety and Efficacy Study of Dose-escalated Hypofractionated Radiotherapy For Prostate Cancer
Acronym: PHART6
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Association of Radiation Oncology (Industry)
Responsible Party: Principal Investigator, Andrew Loblaw, Radiation Oncologist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042-2010
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: Prostatic Neoplasms; Radiotherapy; Hypofractionation; Low and Intermediate Risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT (Experimental): SBRT 40 Gy in 5 fractions over 29 days delivered using step and shoot IGRT
  Interventions: Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 40 Gy / 5 fractions / 29 days

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a short course of radiotherapy (40 Gy / 5 fractions / 29 days) for the treatment of low- and intermediate-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men >18 years
* Histologically confirmed prostate adenocarcinoma
* Low or low-intermediate risk prostate cancer, defined as Clinical stage T1-2b, Gleason Score <=6, and PSA <15 ng/mL, OR Clinical stage T1-2b, Gleason Score 7, and PSA <=10 ng/mL

Exclusion Criteria:

* Prior pelvic radiotherapy
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Presence of a hip prosthesis
* Pelvic girth >40cm - Large prostate (>90cm3) on imaging
* Severe lower urinary tract symptoms (International Prostate Symptom Score >19 or nocturia >3)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 3+ rectal toxicity | Acute period (<3 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v3.0

SECONDARY OUTCOMES:
Incidence of grade 3+ urinary toxicity | Acute (<3 months) and Late (>6 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Quality of Life | 5 years
  Expanded Prostate Cancer Index Composite (EPIC)
Biochemical (ie. prostate specific antigen) disease free survival | 5 year
Incidence of grade 3+ rectal toxicity | Late (>6 months)
  Common Terminology Criteria for Adverse Events (CTCAE) v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Loblaw, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Harvey Quon, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Quon HC, Musunuru HB, Cheung P, Pang G, Mamedov A, D'Alimonte L, Deabreu A, Zhang L, Loblaw A. Dose-Escalated Stereotactic Body Radiation Therapy for Prostate Cancer: Quality-of-Life Comparison of Two Prospective Trials. Front Oncol. 2016 Aug 29;6:185. doi: 10.3389/fonc.2016.00185. eCollection 2016. PMID 27622157